CLINICAL TRIAL: NCT03017196
Title: My Life, My Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Principal Investigator, Kasey R. Boehmer, M.P.H., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-007340
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Sites randomized to intervention will be expected to implement the My Life, My Healthcare Discussion Aid in their practice for at least a 6-month period.
  Interventions: Other: My Life, My Healthcare Discussion Aid
- Control (No Intervention): Sites randomized to control will not be expected to implement the My Life, My Healthcare Discussion Aid in practice. They will be expected to practice chronic care as usual.

INTERVENTIONS:
Other: My Life, My Healthcare Discussion Aid — The My Life, My Healthcare instrument is a conversational tool designed to help patients and clinicians discuss capacity in clinical conversations of primary care.
  Arms: Intervention

SUMMARY:
This study is designed to answer the following questions: "Is the My Life, My Healthcare Discussion Aid feasible for use in primary care? Does it positively impact patient and healthcare teams' care experience and communication, while reducing patient treatment burden?"

Through implementation of the My Life, My Healthcare Discussion Aid for patients with chronic conditions, the study team hypothesizes that it will be feasible to implement in routine primary care practice and positively impact patient and healthcare teams experience of chronic care, while reducing patient treatment burden.

ELIGIBILITY:
InclusionCriteria: Particpant population will include patients 18 years of age or older who have one or more chronic conditions and do not have any barriers to consent (such as major cognitive disabilities) will be eligible for enrollment. Clinicians who treat patients with chronic conditions at participating sites are eligible for enrollment.

Exclusion Criteria: Patients who do not have a chronic condition, or have barriers to consent such as cognitive impairment will be excluded from the study. Health professionals who do not treat patients with chronic conditions will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1929 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Chronic Illness Care (PACIC) | 6 months
  The 20-item scale measures goal setting, coordination of care, decision support, problem solving, and patient activation, and prompts the patient to reflect with items such as: "Over the past 6 months, when I received care for my chronic conditions, I was: helped to make a treatment plan that I could carry out in my daily life."

SECONDARY OUTCOMES:
Illness Intrusiveness Scale | 6 months
  This identifies the extent to which the treatment regimen interferes with life by asking "How much does your illness and/or its treatment interfere with..." things like "your work, including job, house work, chores, or errands?"
General Self-Rated Health | 6 months
  "In general, would you say your health is: Excellent, Very Good, Good, Fair, Poor?"
Communicate with Physician Self-Efficacy Subscale | 6 months
  This 3-item scale has been used in work by Lorig et al. for chronic disease, and asks questions such as "How confident are you that you can discuss openly with your doctor any personal problems that may be related to your illness?"
Consultation Care Measure | 6 months
  This 20-item scale is a valid and discriminating tool to measure communication and partnership, personal relationship, health promotion, positive and clear approach to the problem, and interest in effect of healthcare on patient's life within a single pat
Self-efficacy to Manage Disease in General Subscale | 6 months
  asks questions such as "How confident are you that you can do all the things necessary to manage your condition on a regular basis?"
Treatment Burden Questionnaire (TBQ) | 6 months
  The questionnaire measures the perceived burden of taking medications, self-monitoring and other self-management activities by asking participants to rate the impact of these tasks on a scale from 1-10 with items such as: "The taste, shape or size of your tablets and/or the annoyances caused by your injections (e.g., pain, bleeding, bruising or scars)."
Relational Coordination of Care Team | 6 months
  assesses seven domains of coordinated teams: frequent, timely, accurate, and problem-solving communication, shared goals, shared knowledge, and mutual respect.
Care Team Assessment of Chronic Illness Care (ACIC) | 6 months
  Measures clinician, coach, and clinical team satisfaction with care delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey R. Boehmer, MPH, Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Primary Care Centers of East Kentucky, Hazard, Kentucky
  - Lewis County Primary Care Center, Inc., Vanceburg, Kentucky
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Health System - Springfield, Springfield, Minnesota
  - Vidant Multispecialty Clinic Belhaven, Belhaven, North Carolina
  - Elizabeth Family Medicine, Charlotte, North Carolina
  - CMC- Union Family Medicine, Charlotte, North Carolina
  - Vidant Family Medicine Chocowinity, Chocowinity, North Carolina
  - Mayo Clinic Health System La Crosse, La Crosse, Wisconsin

REFERENCES:
- [Derived] Boehmer KR, Thota A, Organick-Lee P, Branda M, Lee A, Giblon R, Behnken E, Tapp H, May C, Montori V. Care for patients living with chronic conditions using the ICAN Discussion Aid: A mixed methods cluster-randomized trial. PLoS One. 2024 Dec 4;19(12):e0314605. doi: 10.1371/journal.pone.0314605. eCollection 2024. PMID 39630656
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials